CLINICAL TRIAL: NCT03137875
Title: Evaluation of the PCR Using DNA Extracts From Stained Slides and Sputum Collected on Filter Paper for Identification and Detection of Tuberculosis and Multidrug Resistant (MDR) Tuberculosis
Brief Title: Evaluation of PCR Using DNA Extract From Slides and Filter Paper for the Detection of Tuberculosis and MDR-tuberculosis
Status: Completed | Type: Observational
Sponsor: Epicentre (Other)
Collaborators: Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Sponsor
Other Study IDs: HS 918
Record Dates: First submitted 2011-02-22; First posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-04

CONDITIONS: Tuberculosis; Multi Drug Resistant Tuberculosis
Keywords: Tuberculosis; TB; MDR-TB; LIPA; filter paper; slides; MTBDR Plus
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Patient with sputum smear positive 2+: patient who will have a positive diagnostic of tuberculosis using microscopy with a 2+ grade
- patient smear positive scanty or 1+: patient who will have a positive diagnostic of tuberculosis using microscopy with a scanty or 1+ grade
- patient smear negative: patient with a negative TB microscopy result

SUMMARY:
Specimen transport from peripheral health structures to the National TB reference laboratory for MDR-TB identification presents a big challenge in term of sample management, safety, contamination and delays. Thus a system that allows specimen to be collected and shipped in a safely manner while reducing the possibilities of contamination, the cost of shipment and especially the time for detection of MDR-TB by using molecular methods would be very useful. Whereas the some studies show promising results for the development and standardization of simple specimen collection and transportation methods for molecular DST, more data is needed before these can be used in routine.

The study described here aims at identifying a suitable method, in terms of adapted sample support (s) (slide, filter paper (FTA, Genocard ...)) and DNA extraction method. If one or several methods are found to give satisfying results, then a larger patient based evaluation of this (these) method(s) for molecular DST will be performed in a second phase. The protocol for the second phase will be prepared separately.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the performance of PCR in identification and detection of tuberculosis using DNA extracts from stained slides (Ziehl Neelsen and Fluorescence) and Filter paper (FTA card and Genocard).

The secondary objectives of this study are to assess the MTB extraction yield from smear-negative, low and high bacilli load specimens on slides, filter paper ( Genocardand FTA), to determine the amount of sample required to make a detectable PCR reaction and to assess the feasibility of storage and extraction methods.

ELIGIBILITY:
Inclusion Criteria:

* TB suspect with cough more than 2 weeks

Exclusion Criteria:

* None

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will take place in the Mbarara Regional Referral Hospital (MRRH) located in Mbarara Municipality, Mbarara District, and south-west of Uganda.
  Patients suspected of TB are evaluated in the outpatient facility at the hospital or in the medical ward when admitted.
  Some samples will be collected from The Aid Support Organisation (TASO) Mbarara. TASO is located in the neighbourhood of MRRH and EMRB.
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2011-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
proportion of positive samples for Mycobacterium tuberculosis detected by PCR from slides and filter papers among samples by microscopy | 6 MONTHS
  Tests

SECONDARY OUTCOMES:
To assess the MTB extraction yield from smear-negative, low and high bacilli load specimens on slides, filter paper ( Genocardand FTA) | 6 MONTHS
  Tests

CONTACTS AND LOCATIONS:
Overall Officials: Yap JB Boum II, PhD, Study Director — Epicentre Mbarara
Locations (1):
- Epicentre Mbarara Research Base, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No